CLINICAL TRIAL: NCT01374867
Title: Pathophysiology and Prognostic Factors in Cardiogenic Shock - CardShock Study
Brief Title: CardShock Study and Registry
Acronym: CardShock
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Aarne Koskelo Foundation (Other); Finnish Foundation for Cardiovascular Research (Other)
Responsible Party: Principal Investigator, Veli-Pekka Harjola, Chief Physician, Helsinki University Central Hospital
Other Study IDs: 117/13/03/01/2010
Record Dates: First submitted 2011-06-09; First posted 2011-06-16 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2014-01

CONDITIONS: Cardiogenic Shock
Keywords: Cardiogenic shock; Myocardial infarction; Low-output syndrome; Prognosis; Biomarkers; Pathophysiology
MeSH Terms: conditions — Shock, Cardiogenic; Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma, urine
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of CardShock Study is to recognise significant prognostic factors in order to detect patients with increased mortality risk to which one could possibly direct more intensive treatments.

The study will provide clinical, functional and invasive haemodynamic measures with systematic serial sampling and evaluation. In addition, the knowledge on the pathophysiology of cardiogenic shock is increased.

DETAILED DESCRIPTION:
Cardiogenic shock (CS) is a life-threatening emergency situation with high hospital mortality up to 50%. Despite of better treatment strategies including early echocardiography, insertion of pulmonary artery catheter to optimize haemodynamic status, early revascularization therapy, and the use of intra-aortic balloon pump, the prognosis has remained poor and only 50% of patients are discharged alive from the hospital. Most commonly CS occurs after a massive ST-elevation myocardial infarction (AMI) - in 8% of AMIs. The importance of early clinical recognition of the developing CS is the crucial since over 2/3 of CS develop only after hospital admission. In addition, about 20% of the cardiogenic shock patients develop systemic inflammatory response syndrome resembling the clinical picture of septic shock. The clinical picture of CS ranges from florid shock to low-output state. The in-hospital length of stay and the costs of care are many times higher than in other shock or AMI patients

Despite the extreme clinical importance of CS, mostly descriptive parameters but not serial evaluation of biomarkers or clinical condition have been analysed. All in all, the scientific data are still very sparse.

Study design

European investigator initiated multicentre study. A minimum of 100 (up to 200) consecutive patients with cardiogenic shock will be recruited in the study. Standardized treatment protocols of the individual participating centres based on international guidelines on heart failure will be applied to every patient in the study. Coronary angiography with percutaneous coronary intervention, vasoactive and inotropic medication, pulmonary artery catheter and intra-aortic balloon pump are utilized when applicable. Echocardiographies and 14-lead ECG will be recorded. Demographic and clinical data as well as serial blood and urine samples (at up to 8 time points during CCU/ICU stay) are collected.

CardShock Registry The patients who are excluded from the study due to time from onset of shock longer than six hours are recorded to Registry (screening failure) log. These patients will form CardShock Registry which includes clinical data (including in-hospital mortality) but not study sampling nor post-discharge follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Cardiogenic shock with hypotension or severe low output syndrome within 6 hours from identification of it Clinical findings of cardiogenic shock: acute heart failure and

  * Hypotension (systolic blood pressure under 90mmHg despite adequate fluid challenge) over 30 min time
  * OR a need for vasopressor treatment (eg dopamine or norepinephrine) to maintain systolic blood pressure > 90mmHg
  * AND signs of hypoperfusion (either altered mental status, cool periphery, oliguria (< 0.5ml/kg/h for last six hours), or blood lactate > 2 mmol/l)
* Age > 18 years
* Written informed consent by patient or a close person or a relative if the patient is unable to give the consent on admission according to local regulations.

Exclusion Criteria:

* Postoperative patients
* Haemodynamically significant ongoing arrhythmia . (However, e.g. patient resuscitated from serious arrhythmia can be included if the arrhythmia is not ongoing at the time of detection of shock)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2010-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | participants will be followed for 1 year
  during follow-up additional analyses will be performed after ICU/CCU and total hospital stay,and at 90 and 180 days, In patients with impanted cardioverter defibrillator firing for fatal VTach or VFib is recorded
Major cardiac interventions and implantation of devices | 1 year
  Heart transplant, CABG, valve surgery, PCI etc and implantation of devices LVADs, CRT, ICD etc are recorded during follow-up.

SECONDARY OUTCOMES:
Quality of life | 1-year
  The patients will receive EQ5-D questionnaire in their own language and will be asked to fill it at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Veli-Pekka Harjola, MD, PhD, Associate professor, Principal Investigator — Helsinki UCH
Locations (1):
- Helsinki UCH, Helsinki, Finland

REFERENCES:
- [Derived] Liao Y, Luo D, Zhang X, Liu T, Zhang C. Predictive value of age, estimated glomerular filtration rate and ejection fraction (AGEF) score for all-cause 90-day mortality in patients with cardiogenic shock. J Cardiovasc Med (Hagerstown). 2025 Jun 1;26(6):269-279. doi: 10.2459/JCM.0000000000001729. Epub 2025 May 2. PMID 40472170
- [Derived] Jantti T, Tarvasmaki T, Harjola VP, Pulkki K, Turkia H, Sabell T, Tolppanen H, Jurkko R, Hongisto M, Kataja A, Sionis A, Silva-Cardoso J, Banaszewski M, DiSomma S, Mebazaa A, Haapio M, Lassus J; CardShock investigators. Predictive value of plasma proenkephalin and neutrophil gelatinase-associated lipocalin in acute kidney injury and mortality in cardiogenic shock. Ann Intensive Care. 2021 Feb 5;11(1):25. doi: 10.1186/s13613-021-00814-8. PMID 33547528
- [Derived] Jantti T, Tarvasmaki T, Harjola VP, Parissis J, Pulkki K, Javanainen T, Tolppanen H, Jurkko R, Hongisto M, Kataja A, Sionis A, Silva-Cardoso J, Banaszewski M, Spinar J, Mebazaa A, Lassus J; CardShock investigators. Hypoalbuminemia is a frequent marker of increased mortality in cardiogenic shock. PLoS One. 2019 May 16;14(5):e0217006. doi: 10.1371/journal.pone.0217006. eCollection 2019. PMID 31095609
- [Derived] Tolppanen H, Rivas-Lasarte M, Lassus J, Sadoune M, Gayat E, Pulkki K, Arrigo M, Krastinova E, Sionis A, Parissis J, Spinar J, Januzzi J, Harjola VP, Mebazaa A; CardShock Investigators. Combined Measurement of Soluble ST2 and Amino-Terminal Pro-B-Type Natriuretic Peptide Provides Early Assessment of Severity in Cardiogenic Shock Complicating Acute Coronary Syndrome. Crit Care Med. 2017 Jul;45(7):e666-e673. doi: 10.1097/CCM.0000000000002336. PMID 28403119
- [Derived] Tolppanen H, Rivas-Lasarte M, Lassus J, Sans-Rosello J, Hartmann O, Lindholm M, Arrigo M, Tarvasmaki T, Kober L, Thiele H, Pulkki K, Spinar J, Parissis J, Banaszewski M, Silva-Cardoso J, Carubelli V, Sionis A, Harjola VP, Mebazaa A. Adrenomedullin: a marker of impaired hemodynamics, organ dysfunction, and poor prognosis in cardiogenic shock. Ann Intensive Care. 2017 Dec;7(1):6. doi: 10.1186/s13613-016-0229-2. Epub 2017 Jan 4. PMID 28050899
- [Derived] Harjola VP, Lassus J, Sionis A, Kober L, Tarvasmaki T, Spinar J, Parissis J, Banaszewski M, Silva-Cardoso J, Carubelli V, Di Somma S, Tolppanen H, Zeymer U, Thiele H, Nieminen MS, Mebazaa A; CardShock Study Investigators; GREAT network. Clinical picture and risk prediction of short-term mortality in cardiogenic shock. Eur J Heart Fail. 2015 May;17(5):501-9. doi: 10.1002/ejhf.260. Epub 2015 Mar 28. PMID 25820680